CLINICAL TRIAL: NCT02914028
Title: Evaluation of the Effects of Subcostal Transversus Abdominis Plane Block on Subacute Pain Development Following Inguinal Herniography: a Randomized Clinical Study
Brief Title: TAP Block and Subacute Pain in Inguinal Herniography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr Cigdem Akyol Beyoğlu, medical doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 235901
Record Dates: First submitted 2016-08-26; First posted 2016-09-26 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain
Keywords: TAP block; subacute pain; inguinal herniography
MeSH Terms: conditions — Pain, Postoperative | interventions — Ultracet; Tramadol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol and paracetamol (Active Comparator): subjects were administered intravenous analgesia (control group) Tramadol 100 mg and paracetamol 1000 mg at the end of the surgery
  Interventions: Drug: Tramadol and paracetamol
- transversus abdominis plane block (Active Comparator): patients that applied transversus abdominis plane block at the end of the surgery after given intravenous analgesia
  Interventions: Procedure: transversus abdominis plane block; Drug: Tramadol and paracetamol

INTERVENTIONS:
Procedure: transversus abdominis plane block — A peripheric block needle is inserted entering the facia between musculus rectus abdominis and musculus transversus abdominis with ultrasonography and local anesthetics are injected in the facia.
  Other Names: stimuplex A
  Arms: transversus abdominis plane block
Drug: Tramadol and paracetamol — Tramadol 100 mg and paracetamol 1000 mg are applied to the patients at the end of the surgery
  Other Names: contramal; parol infusion solution

SUMMARY:
Inguinal hernia repair with mesh has a high incidence of postoperative chronic pain. Transversus abdominis plane block is a current intervention to support postoperative analgesia, however it is recently in research area how to be applied in different surgical areas to be more effective than intravenous opioids. Subcostal transversus abdominis plane block is not advised but has not been studied to be effective for postoperative analgesia in inguinal herniography patients.

This study aims to research the effect of subcostal transversus abdominis plane block in subacute postoperative pain after inguinal hernia repair

DETAILED DESCRIPTION:
Patients were divided into two groups, one is control and the second is subcostal transversus abdominis plane block (STAP) group. After standard general anesthesia application, control group ( Group I) had 1 gram of paracetamol and 100 mg of contramal just after starting surgical closure. Group II (STAP) had 1 gram of paracetamol and 100 mg of contramal, after surgical closure transversus abdominis plane block in subcostal area was applied to the patient.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* who were to undergo elective unilateral inguinal herniography with "mesh" under general anesthesia.

Exclusion Criteria:

* patients who have allergy to local anesthetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
verbal numeric scale | 1 month after the operation
  patients were questioned for pain graduation to give a point from 0 to 10 according to the intensity of the pain. 0 equals to no pain, 10 equals to the strongest pain

SECONDARY OUTCOMES:
verbal numeric scale | 15 minutes, 1-6-12-24 hours and 15 days after operation
  according to the intensity of the pain. 0 equals to no pain, 10 equals to the strongest pain

IPD SHARING:
Plan to Share IPD: No